CLINICAL TRIAL: NCT03473028
Title: Could Transvaginal Ultrasonography Guided Embryo Transfer Improves Pregnancy Outcome in Obese Patients Undergoing Intracytoplasmic Sperm Inoculation? Randomized Controlled Study
Brief Title: Transvaginal Ultrasonography Guided Embryo Transfer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, sarah mohamed hassan, lecturer of obstetrics and gynecology, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019
Record Dates: First submitted 2018-03-15; First posted 2018-03-21 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Infertility, Female
Keywords: obesity; embryo transfer; invitro fertilization
MeSH Terms: conditions — Infertility, Female; Obesity

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transabdominal ultrasound (Active Comparator): 400 obese female undergo transabdominal ultrasound guided embryo transfer
  Interventions: Procedure: transabdominal ultrasound guided embryo transfer
- transvaginal group (Active Comparator): 400 obese female undergo transvaginal ultrasound guided embryo transfer
  Interventions: Procedure: transvaginal ultrasound guided embryo transfer

INTERVENTIONS:
Procedure: transabdominal ultrasound guided embryo transfer — 400 female with body mass index more than 30undergo transabdominal ultrasound guided embryo transfer
  Arms: transabdominal ultrasound
Procedure: transvaginal ultrasound guided embryo transfer — 400 female with body mass index more than 30 undergo transvaginal ultrasound guided embryo transfer
  Arms: transvaginal group

SUMMARY:
to evaluate the value of using transvaginal ultrasound guided embryo transfer in obese patients undergoing in vitro fertilization.

DETAILED DESCRIPTION:
The 800 participants with body mass index more than 30kg/m2 were randomly allocated to two groups of equal size using an automated web-based randomization system. The first group 400 patient undergoing the transabdominal-guided embryo transfer, the second group 400 patient undergoing transvaginal-guided embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* BMI more than 35, good ovarian reserve, unexplained infertility more than 3 years.

Exclusion Criteria:

* severe male factor of infertility,uterine factor of infertility excluded by ultrasonography and hysteroscopy ,ovarian endometrioma or patients with poly cystic ovary syndrome, obesity caused by abnormal endocrine function (thyroid or adrenal disorder)

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 800 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate' | 4 weeks following embryo transfer
  the presence of at least one intrauterine gestational sac with viable fetus.

SECONDARY OUTCOMES:
live birth rate | immediately following delivery
  delivery of a living baby

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Ainiy Hospital, Cairo, Egypt

REFERENCES:
- [Derived] Mohamed Hassan S, Ramadan W, Elsharkawy M, Ali Bayoumi Y. The Role of Transvaginal Ultrasound Guided Embryo Transfer to Improve Pregnancy Rate in Obese Patients Undergoing Intracytoplasmic Sperm Injection. Int J Womens Health. 2021 Sep 21;13:861-867. doi: 10.2147/IJWH.S325557. eCollection 2021. PMID 34584462